CLINICAL TRIAL: NCT06063434
Title: Testing the Effectiveness of a Theory-based, Customized Video Game at Increasing the Implementation of Clinical Practice Guidelines in Trauma Triage
Brief Title: Testing the Effectiveness of Night Shift, a Theory-based Customized Video Game
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Deepika Mohan, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY23070156; R01AG076499 (NIH)
Record Dates: First submitted 2023-09-20; First posted 2023-10-02 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Trauma Injury; Physician's Role
Keywords: Heuristics; Serious game; Guidelines
MeSH Terms: conditions — Accidental Injuries | interventions — Shift Work Schedule

STUDY DESIGN:
Intervention Model Description: Physicians will be randomized in a 1:1 fashion to the intervention condition or to the control condition.
Who Masked: Outcomes Assessor
Masking Description: Participant assignment will be masked within the data with unblinding occurring only after data cleaning has completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Night Shift (Experimental): Night Shift 2024 is a customized, theory-based adventure video game in which the player takes on the character of Andy Jordan, a young emergency medicine physician who moves home after the disappearance of his grandfather and takes a job at a local community hospital. The investigators will ask participants to play Night Shift for 2 hours upon enrollment (or within 2 weeks), and then come back to the game quarterly to play it again for 20 minute booster sessions. They will unlock additional game content each quarter to make the experience more enjoyable.
  Interventions: Behavioral: Night Shift
- Usual education (Active Comparator): Participants will receive their usual continuing medical education, but nothing additional.
  Interventions: Behavioral: Usual education

INTERVENTIONS:
Behavioral: Night Shift — The player must not only manage the patients who present to the emergency department of the hospital, gaining experience with the consequences of trauma triage, but also solve the mystery of the grandfather, gaining an emotional connection with the character and making the feedback that "Andy" receives more relevant. Embedded within Night Shift 2024 is a mini-game (Graveyard Shift) that contains a series of puzzles that reinforce the lessons of the overarching game: transfer severely injured patients expeditiously.
  Arms: Night Shift
Behavioral: Usual education — Standard continuing medical education, including Advanced Trauma Life Support, and the American Board of Emergency Medicine educational modules (e.g., trauma resuscitation).
  Arms: Usual education

SUMMARY:
The goal of this clinical trial is to test the effect of a video game on the implementation of clinical practice guidelines in trauma triage. The main question it attempts to answer is whether exposure to the game improves compliance with guidelines by emergency medicine physicians working at non-trauma centers in the US. Participants randomized to the intervention condition will be asked to play a customized, theory-based video game for 2 hours immediately after enrollment, and then return to the game for 20 minutes every three months for the next 9 months. Participants in the control condition will receive usual care.

DETAILED DESCRIPTION:
Transfer of severely injured patients to trauma centers, either directly from the field or after evaluation at non-trauma centers, reduces preventable morbidity and mortality. Failure to transfer these patients appropriately (i.e., under-triage) remains common, and occurs in part because physicians at non-trauma centers make diagnostic errors when evaluating the severity of patients' injuries. The study team developed Night Shift, a theory-based adventure video game, to recalibrate physician heuristics (intuitive judgments) in trauma triage and established its efficacy in the laboratory. The investigators plan a Type 1 hybrid effectiveness-implementation trial to determine whether the game changes physician triage decisions in real-life, and hypothesize that it will reduce the proportion of patients under-triaged.

ELIGIBILITY:
Inclusion Criteria:

- Board certified physicians who work exclusively in the emergency departments (EDs) of non-trauma centers in the US AND triage adult trauma patients

Exclusion Criteria:

* non-physician healthcare professionals who work in EDs
* physicians who work at trauma and non-trauma centers
* physicians who work outside the continental US

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Under-triage | 1 year
  Proportion of severely injured patients, treated by trial participants, not transferred to a higher level of care after initial evaluation at a non-trauma center

SECONDARY OUTCOMES:
Mortality and hospital readmission | 1 year
  Proportion of severely injured patients, treated by trial participants, who die or are readmitted to any hospital within 30 days of their initial evaluation at a non-trauma center
Functional dependence | 1 year
  Proportion of severely injured patients, treated by trial participants, with 90-day preadmission location at home with discharge to a skilled nursing or rehabilitation facility after initial treatment at a non-trauma center.
Over-triage | 1 year
  Proportion of injured patients, treated by trial participants, transferred to a higher level of care after initial evaluation at a non-trauma center with minimal injuries

CONTACTS AND LOCATIONS:
Overall Officials: Deepika Mohan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The protocol, primary data, and meta-data (e.g., documentation, protocols used to clean and to manage the data), will be uploaded to the open access Inter-university Consortium for Political and Social Research (open ICPSR) repository at the conclusion of the trial. Of note, data obtained from Medicare will not be shared as part of the results of the trial, because we do not own those records.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 6 months after publication of the primary manuscript.
Access Criteria: We will upload the data to the open ICPSR repository, where other researchers can access it.

REFERENCES:
- [Derived] Mohan D, Fischhoff B, Talisa V, Elmer J, White DB, Angus DC, Peitzman A, Bendesky B, Chapman AC, Forsythe RM, Guyette FX, Hynes AM, Oskvarek JJ, Weingart SD, Weinstock M, Chang CH. An Educational Video Game in Trauma Triage at Nontrauma Centers: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Jun 2;8(6):e2513375. doi: 10.1001/jamanetworkopen.2025.13375. PMID 40465299
- [Derived] Mohan D, Angus DC, Chang CH, Elmer J, Fischhoff B, Rak KJ, Barnes JL, Peitzman AB, White DB. Using a theory-based, customized video game as an educational tool to improve physicians' trauma triage decisions: study protocol for a randomized cluster trial. Trials. 2024 Feb 16;25(1):127. doi: 10.1186/s13063-024-07961-w. PMID 38365758

DOCUMENTS (1):
  • Informed Consent Form (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT06063434/ICF_000.pdf